CLINICAL TRIAL: NCT02259452
Title: Radiation Induced Cardiopulmonary Injury in Humans
Status: Terminated | Type: Observational
Why Stopped: Decision to not gather further data
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC0808
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Thoracic; Pulmonary Injury; Heart Injuries
Keywords: Radiation Therapy
MeSH Terms: conditions — Lung Injury; Heart Injuries | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: SPECT Lung Perfusion Scan
Procedure: SPECT Heart Perfusion Scan
Procedure: Pulmonary Function Tests

SUMMARY:
The purpose of the study is to assess the time, dose dependence, and fraction-size dependence of radiation (RT)-induced changes in regional lung and heart perfusion/function/structure following thoracic RT delivered using newer IMRT/conformal/radiosurgery techniques. The PI hopes to develop models to better relate and predict RT-induced changes in regional lung and heart perfusion/function/structure with changes in global cardiopulmonary function. Patients will undergo pre- and serial post-RT lung and heart assessments to better understand RT-induced regional heart/lung changes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients who are to receive 3D-planned RT for tumor within and around the thorax.
3. Patients receiving incidental RT to portions of the heart are eligible.
4. Estimated minimum expected life expectancy of one year
5. Able to undergo the required study-related tests for regional lung injury and regional heart injury
6. Patients of child bearing potential age must have a negative pregnancy test and must agree to use appropriate birth control measures while in the study.
7. Patients must be able to give informed consent. Informed consent will be obtained prior to enrollment.

Exclusion Criteria:

1. Patients who are anticipated to have thoracic surgery post-RT are ineligible.
2. Patients with large mediastinal/hilar tumors compressing the airways/vessels, and negatively impacting on cardiovascular function
3. Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are to receive 3D-planned RT for lung cancer (conformal or IMRT) or other tumors in/around the thorax.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2008-06; Primary Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Changes in Regional Lung Function | Up to 4 years post CRT
Changes in Regional Heart Function | Up to 4 years post CRT
Relating RT-Induced Changes in Regional injury to Global Cardiopulmonary Changes | Up to 4 years post CRT

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Wang, MD, Principal Investigator — University of North Carolina at Chapel Hill, Department of Radiation Oncology
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States